CLINICAL TRIAL: NCT00907010
Title: Sarcopenia and Aging
Status: Completed | Type: Observational
Sponsor: Universidade de Franca (Other)
Responsible Party: Lislei Jorge Patrizzi, Universidade de Franca
Other Study IDs: 088/08; 088/08
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Sarcopenia
Keywords: Ageing; Sarcopenia; Muscular contraction
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Biospecimen Retention: The evaluation instruments used were: (1) Esfigmomanômetro (EM), (2) Trunk flexor in the supine position,, (3) Jamar Dinamômetro and (4) Preston Pinch Gauge Dinamômetro.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I: 11 to 18 years - composed of 12 adolescent with six women and six men
- Group II: 20 to 26 years - composed of 12 young with six women and six men
- Group III: 45 to 60 years - composed of 12 adult with six women and six men
- Group IV: 66 - 82 years - composed of 12 aged with six women and six men

SUMMARY:
Objective: Evaluate the muscular strength in the ageing process and identify the changes between the abdominal muscles, upper and louver edges.

Method: 48 individuals participated in this study, being divided into four groups according to the age: (G1) 11to 18 years old, (G2) 20 to 26 years old, (G3) 45 to 60 years old and (G4) 66 - 82 years old. The excluding criterion included people who work out more than three times a week, severe arthrosin, stroke, significant cognitive deficit , obesity, use of ortheses for louver members or any break, with or without metallic implant. The evaluation instruments used were: (1) Esfigmomanômetro (EM), (2) Trunk flexor in the supine position,, (3) Jamar Dinamômetro and (4) Preston Pinch Gauge Dinamômetro.

DETAILED DESCRIPTION:
Forty-eight subjects participated voluntarily in this work and is divided into four groups of 12 participants with 6 men and 6 women: (G1) 11 to 18 years (G2) 20 to 26 years (G3) from 45 to 60 and (G4) 66 to 82 years, selected in dependency of Unifran and residences of the city of Franca, Sao Paulo - Brazil. To evaluate muscle strength, a BD sphygmomanometer was used to analyze the strength of flexors and extensors of the knee. The Jamar Dynamometer was used to assess the functional integrity of the upper and Preston Pinch Gauge Dynamometer for evaluation of gripper hands.

ELIGIBILITY:
Inclusion Criteria:

* absence of the basic pathology that interferes directly in the muscle

Exclusion Criteria:

* people who work out more than three times a week
* severe arthrosin
* stroke
* significant cognitive deficit
* obesity
* use of ortheses for louver members or any break
* with or without metallic implant

Ages: 11 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 48 individuals participated in this study, being divided into four groups according to the age: (G1) 11to 18 years old, (G2) 20 to 26 years old, (G3) 45 to 60 years old and (G4) 66 - 82 years old.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lislei Patrizzi, Study Director — Universidade de Franca